CLINICAL TRIAL: NCT07139106
Title: Dynorphin/Kappa Opioid Receptor Signaling Role in Ketamine's Anti-suicidal Ideation Effect
Brief Title: Understanding the Role of the Kappa Opioid Receptor in Ketamine's Attenuation of Suicidal Thoughts
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Elizabeth Bartlett, Assistant Professor of Clinical Neurobiology in Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00089428; ECR-0-013-24 (Other Grant/Funding Number: American Foundation for Suicide Prevention)
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: ketamine; positron emission tomography (PET); kappa opioid receptor; major depressive disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine (Experimental): single racemic ketamine hydrochloride 0.5 mg/kg infusion
  Interventions: Drug: Ketamine hydrochloride infusion

INTERVENTIONS:
Drug: Ketamine hydrochloride infusion — single racemic ketamine hydrochloride 0.5 mg/kg infusion

SUMMARY:
This study explores how stress, suicidal thoughts, and ketamine's effects are connected in people with major depressive disorder. Stress increases the risk for suicidal thoughts, but the biological basis is unclear. Ketamine may help reduce suicidal thoughts by affecting stress-linked brain systems. This study will use smartphone tracking to monitor real-time responses to stress and positron emission tomography (PET) brain scans to study how ketamine affects brain pathways related to stress and suicidal thoughts in depressed individuals.

ELIGIBILITY:
Inclusion Criteria:

* DSM5 unipolar major depressive episode
* Persons of child-bearing potential must agree to use an acceptable method of birth control throughout the study.

Exclusion Criteria:

* Current or past ketamine abuse or dependence ever (lifetime)
* Any medical contraindication to ketamine, including prior ineffective trial of or medically significant adverse reaction to ketamine.
* Clinically significant EKG abnormality in terms of ketamine administration (e.g., Ventricular tachycardia, evidence of myocardial ischemia, symptomatic bradycardia, unstable tachycardia, second degree (or greater) AV block).
* Lifetime schizophrenia, schizoaffective illness, bipolar disorder, current psychotic depression; mild drug or alcohol use disorder in past 2 months; moderate or severe drug or alcohol use disorder in past 6 months; suicidal ideation with plan and/or intent within 6 months; suicide attempt in the past month.
* A first-degree family history of schizophrenia if the subject is less than 33 years old (mean age of onset for schizophrenia plus two standard deviations).
* Current or recent use of antidepressants within 14 days or benzodiazepines within 1 day. Use of fluoxetine or other long-acting antidepressant within 6 weeks.
* Current or recent use of medications known to affect brain biology of interest such as competing for binding sites of PET tracer within 1 month.
* Uncontrolled moderate or severe hypertension (≥160 mmHg systolic or ≥100 mmHg diastolic[41]), history of Raynaud's phenomenon, seizures, an open cut, sore, or bone fracture on or near the hands to be used for the cold pressor test.
* Use of more than incidental NSAIDs (including aspirin), anti-inflammatories, immune suppressants or other pain medications.
* Significant active physical illness, particularly if it may affect the brain biology being studied; including chronic pain syndrome and medically compromising eating disorders or epilepsy.
* Lacks capacity to consent
* Aggressive behavior that is a significant threat to others such as physically assaultive behavior (in the last month).
* Pregnancy, abortion or miscarriage in the previous two months or plans to conceive during the course of study participation.
* Currently lactating
* Previous head injury with evidence of cognitive impairment. Subjects who endorse a history of prior head trauma and score 1.5 standard deviations below the mean on Trail-making A or B will be excluded from study participation.
* Any condition or material in the body that is a contraindication for MRI procedures.
* Current, past or anticipated exposure to radiation except if the exposure was at our PET center where the precise exposure is known
* ECT within past 6 months
* For A-Line Subjects: Unstable relevant medical condition (i.e., condition not adequately stabilized for 3 months). Including bleeding disorders, the need to take medications that affect blood clotting, and certain platelet and hemoglobin cutoffs
* Blind or with visual impairment that cannot be corrected with corrective lenses (glasses or contact lenses)
* No emergency contact

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Scale for Suicidal Ideation (SSI) | 24 hours post-treatment
  Beck Scale for Suicidal Ideation clinician-rated version. Minimum score = 0, Maximum score = 38. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All associated research findings published will be made readily available for research purposes to qualified individuals within the scientific community. All data will be made anonymous (de-identified) and available after written requests for data are submitted by such qualified individuals to the PI.